CLINICAL TRIAL: NCT03797105
Title: Frequency of Intervention Needed to Improve Weight Outcomes of Mexican-American Adolescents With Overweight or Obesity
Brief Title: Frequency Needed for School-based Obesity Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Craig A Johnston, Associate Professor, University of Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000487
Record Dates: First submitted 2019-01-04; First posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Obesity, Child
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control, 0 days (No Intervention): control group, no intervention
- 1 day (Experimental): received the intervention 1 day/week
  Interventions: Behavioral: School-Based Obesity Intervention (FLOW)
- 3 days (Experimental): received the intervention 3 days/week
  Interventions: Behavioral: School-Based Obesity Intervention (FLOW)
- 5 days (Experimental): received the intervention 5 days/week
  Interventions: Behavioral: School-Based Obesity Intervention (FLOW)

INTERVENTIONS:
Behavioral: School-Based Obesity Intervention (FLOW) — The intervention consisted of nutrition lessons based on the traffic light diet, circuit-based physical activity, behavior modification techniques (token economy system, goal setting, self-monitoring), and parental involvement (materials sent home and monthly parent meetings). 80% of time was spent on physical activity and 20% was spent on nutrition. Behavior modification was incorporated into both physical activity and nutrition time. Specifically, instruction and activity time during PE class lasted approximately 40 minutes.
  Arms: 1 day; 3 days; 5 days

SUMMARY:
This randomized controlled trial compared changes in Mexican-American, adolescent standardized body mass index (zBMI) from a school-based obesity intervention given zero, one, three, or five days a week.

DETAILED DESCRIPTION:
Efficacious school-based interventions have been intensive making it difficult for interventions to be scaled. The more components there are to an intervention, typically the better the results. Instead of decreasing intensity via the removal of intervention components, this randomized controlled trial aimed to compare changes in Mexican-American adolescent standardized body mass index (zBMI) based on the number of days per week they received a multi-component intervention. Mexican-American middle school students (n=203) with overweight or obesity were recruited from an independent school district in Houston. Students were randomized to receive an obesity intervention with established efficacy zero (control), one, three, or five days/week. In each condition, 80% of intervention time was allocated to physical activity and 20% to nutrition. Directly measured height and weight were used to calculate zBMI.

ELIGIBILITY:
Inclusion Criteria:

1. BMI-for-age (Body Mass Index) percentile ≥ 85
2. Male or female between ages 10 - 17 years
3. Self-identified as Mexican-American

Exclusion Criteria:

1. Student who is pregnant, planning to become pregnant, or becomes pregnant
2. School report of cognitive impairment significantly below average age and/or grade level
3. Use of any weight-loss medication (prescription or nonprescription) for at least 6 months prior to screening
4. Type 1 or 2 diabetes medical diagnosis

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 243 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2014-09-30 (Actual); Study Completion 2014-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Standardized Body Mass Index (zBMI) | baseline, 6, and 12 months
  standardized body mass index

CONTACTS AND LOCATIONS:
Overall Officials: Craig A Johnston, PhD, Principal Investigator — University of Houston
Locations (1):
- YES Prep Brays Oaks, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers